CLINICAL TRIAL: NCT01208948
Title: Alpha Lipoic Acid in the Treatment of Diabetic Retinopathy
Brief Title: Clinical Trial on Alpha Lipoic Acid in Diabetic Macular Edema
Acronym: RETIPON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Prof. Dr. Anselm Kampik, Ludwig-Maximilians-University, Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DMP 77.1.99
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus; Macular Edema
Keywords: macular edema; diabetes mellitus; prevention alpha lipoic acid
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alpha lipoic acid 600 mg (Active Comparator)
  Interventions: Drug: 1,2 dithiolane 3 valeric acid
- placebo pill (Placebo Comparator)
  Interventions: Drug: 1,2 dithiolane 3 valeric acid

INTERVENTIONS:
Drug: 1,2 dithiolane 3 valeric acid — 600 mg alpha lipoic acid per day

SUMMARY:
To evaluate the effect of alpha lipoic acid (ALA) on the occurrence of diabetic macular edema.

DETAILED DESCRIPTION:
Randomised, double-blind, placebo controlled multicentre study. Patients were randomised to the treatment group with 600 mg ALA per day or the placebo group. At each examination we took stereo fundus photographs, HbA1c levels, and performed an ophthalmological examination. Primary endpoint of the study was the occurrence of clinically significant macular edema (CSME) within a follow-up period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type II, mild non proliferative diabetic retinopathy,
* Microalbuminuria > 30 mg/L

Exclusion Criteria:

Ophthalmic exclusion criteria

* severe non-proliferative or proliferative diabetic retinopathy
* Macular edema
* Eye diseases interfering with the examinations of the fundus such as preretinal haemorrhage, cataract, vitreous haemorrhage
* Amblyopia
* Best corrected visual acuity (VA) over 0.5
* Glaucoma
* Patients with cataract surgery within a period of three months
* Other relevant retinal diseases
* Non-authorized interventional therapy of diabetic retinopathy (e.g. laser, kryo-coagulation, vitrectomy)
* General exclusion criteria
* Chronic administration of alpha lipoic acid or of more than five successive days during the last twelve months
* Known intolerance/hypersensitivity to alpha lipoic acid
* Type I diabetes mellitus
* Poor metabolic control with HbA1c >10.5 %/dl
* Late sequelae of diabetes with organic manifestation (e.g. dialysis in cases of renal insufficiency, history of kidney transplantation, creatinine > 1.6 mg/dl)
* Poorly controlled arterial hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 95 mmHg)
* Severe disturbances in lipid metabolism (triglycerides > 500 mg/dl or total cholesterol > 320 mg/dl)
* Unpermitted concomitant medication defined as any medicine with a potential interaction with alpha lipoic acid or with the effect of alpha lipoic acid were excluded as concomitant medication. These included aldose reductase inhibitors, substances promoting blood flow, anticoagulants apart from acetylsalicylic acid 500 mg/day and short-term treatment of diseases with the normal dose of acetylsalicylic acid, chronically and systemically administered corticosteroids, hormonal contraceptives
* Malignancies or life threatening diseases
* Drug or alcohol abuse
* Blood donation or blood loss greater than 500 ml) within the last 3 months
* Pregnancy or breast feeding
* Participation in a clinical trial within the last 30 days

Ages: 45 Years to 68 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2000-07; Primary Completion 2005-04 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
occurrence of clinically significant macular edema (CSME) within a follow-up period of 2 years | two years

SECONDARY OUTCOMES:
The time to CSME development | two years

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Ulbig, MD, Study Director — Ludwig-Maximilians - University of Munich
Locations (1):
- Department of Ophthalmology, Munich, Germany, Germany